CLINICAL TRIAL: NCT01764607
Title: A Phase II Study of Sirolimus in Renal Transplant Patients Diagnosed With New or Recurrent Squamous Cell Skin Carcinoma Currently on Calcineurin-based Immunosuppression.
Brief Title: Sirolimus in Kidney Transplant Patients With Squamous Cell Skin Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 514-2012; 00086505 (Other Grant/Funding Number: University of Florida)
Record Dates: First submitted 2012-12-18; First posted 2013-01-09 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Squamous Cell Skin Carcinoma
Keywords: Squamous; Renal; Transplant
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus treatment (Experimental): Patients will receive sirolimus 5 weeks prior to removal of squamous cell skin carcinoma. After the 5 weeks of treatment, nephrology will determine/manage each patient's immunosuppressant therapy.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Patients randomized to this arm of the study will receive sirolimus from the time of randomization at least until 5 weeks or the removal of the skin tumor. Nephrology will determine/manage the immunosuppressant therapy.
  Other Names: Rapamune

SUMMARY:
Solid organ transplant recipients (SOTR) have a 3-5x increased occurrence of cancer in contrast to the general population with basal and squamous cell skin cancer. The use of immunosuppressant or anti-rejection drugs that are needed after SOTR is known to increase the risk of developing certain kinds of cancer. The purpose of this study is to find out how well Sirolimus (also known as Rapamune) works at treating squamous cell carcinoma in renal transplant patients.

DETAILED DESCRIPTION:
This is a Phase II randomized study to evaluate the effectiveness of Sirolimus in treating and preventing squamous cell skin cancer carcinoma using a Simon's 2-stage design. As part of the study, after the biopsy results of the skin cancer show squamous cell carcinoma and consent had been obtain, the participant will begin taking Sirolimus. The calcineurin inhibitor (tacrolimus or cyclosporine) will be discontinued once the transplant doctors find that the participants Sirolimus is therapeutic by checking blood tests once a week x 3 weeks. Approximately 5 weeks after starting Sirolimus, the squamous cell skin cancer will be removed by a surgeon. Participant next follow up visit for the study is scheduled one year post-operatively. .The study will look at your squamous cell skin cancer under the microscope to see if sirolimus had any effect at treating your squamous cell skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell skin carcinoma
* Recipient of a renal organ transplant at least one year prior to study enrollment
* Receiving a CNI for at least 6 months prior to diagnosis of skin cancer
* No current evidence of graft rejection, except low-grade, chronic graft rejection
* Measurable disease by caliper measurement
* Life expectancy > 6 months
* Age of at least 18 years
* Adequate organ and marrow function as determined by ANC, HGB, PLT, Total Bili, AST, and creatinine clearance
* Ability to understand/willingness to sign a written informed consent form

Exclusion Criteria:

* Inability to give informed consent
* Major surgery within 4 week prior to starting study drug
* Chronic or non-healing open wounds
* Pregnant and nursing women
* Women and men of child-bearing potential must agree to use adequate contraception prior to study entry and for the study duration
* Prior use of an mTOR inhibitor
* Pre-existing clinically significant cardiac, hepatic, pulmonary, or renal dysfunction
* HIV-positive patients
* Proteinuria (> 1 gram)
* Prior or current history of uncontrolled hyperlipidemia (cholesterol > 302 mg/dl or triglycerides 354 mg/dl
* Currently receiving any investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sirolimus (mTOR inhibitors)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Gopalan, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure of Squamous Cell Skin Carcinoma in Patients
Description: Baseline: Measuring of squamous cell skin carcinoma, Week 5: Measuring and surgical removal of squamous cell skin cancer with microscopic evaluation, and in 1 year.
Time Frame: Baseline, time of surgical removal (5 weeks) and 1 year.
Measure: Number; unit: mm
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 1
mm
  Measurement at Baseline | 15
  Measurement at 5 Weeks | 12
  Measurement at 1 Year | 0

2. Secondary Outcome: Evaluation of Skin Tumor for Squamous Cell Skin Carcinoma
Description: Tumor will be analyzed at baseline and time of surgical removal by both laboratory and microscopic testing.
Time Frame: At baseline and time of surgical removal (5 weeks).
Measure: Number; unit: percentage of baseline size
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 1
percentage of baseline size | 80

ADVERSE EVENTS:
Arm/Group | Sirolimus Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Treatment (N=1)
Hypertension (Cardiac disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No